CLINICAL TRIAL: NCT00836771
Title: Evaluation of the Effect of Milk Based Infant Formula Supplemented Either With Probiotic Microorganisms and/or With Prebiotic on the Intestinal Microflora During the First 4 Months of Life of Healthy, Full Term Infants and it's Long Term Effect on Morbidity up to the Age of 9 Months
Brief Title: Infant Formula Supplemented With Probiotic Microorganisms and/or Prebiotic.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Materna Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 80801
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2012-05

CONDITIONS: Focus on Healthy Infant Growth.
Keywords: Infant formula; Probiotic microorganisms; prebiotic
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Materna infant formula 1 (Placebo Comparator): milk based infant formula powder
  Interventions: Dietary Supplement: Infant Formula
- Materna infant formula 2 (Experimental): Probiotic supplemented infant formula
  Interventions: Dietary Supplement: Infant Formula
- Materna infant formula 3 (Experimental): Prebiotic supplemented infant formula
  Interventions: Dietary Supplement: Infant Formula
- Materna infant formula 4 (Experimental): Prebiotic+ Probiotic supplemented infant formula
  Interventions: Dietary Supplement: Infant Formula
- Human milk (Other): Human Milk
  Interventions: Dietary Supplement: Infant Formula

INTERVENTIONS:
Dietary Supplement: Infant Formula
  Other Names: Materna

SUMMARY:
Evaluation the nutritional suitability of a based milk infant formula supplemented with friendly bacteria (probiotic microorganisms) and or nutritional fibers (prebiotic) to healthy, full term infants compare with an otherwise identical widely used commercially available milk based infant formula and/or breast feed

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants of both sexes, born in natural labor .
* Single birth.
* Full term infants (born between the 37th and 42nd week of gestation)
* Infants with birth weight >2500 g.
* Recruitment age will be 0-21 days.
* Infants whose mothers are unable to breast feed or have chosen not to breast feed prior to the study enrollment.
* Infants whose parents have agreed to participate in the study up to the age of 9 months..
* Infants whose parents have agreed to remain exclusively on the same product for 16 weeks of age..
* Infants whose parents have signed the informed consent form.
* Infants whose parents are able to understand the protocol requirements and to fill out the infant's diary and agree to completely fill out the parents' questionnaires during the period Of 9 months

Exclusion Criteria:

* Twins.
* Premature or low birth weight (< 2500 g).
* Chromosomal abnormalities or congenital malformation.
* Suffering jaundice which require phototherapy.
* Proven or suspected family history of allergy to cow's milk.
* Having been treated with antibiotics or other drugs during the last three days or more prior to the commencement of the study.

Ages: 1 Day to 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 270 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-01 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
weight gain | 1 to 120 days of age

SECONDARY OUTCOMES:
Anthropometric | 1-120 days of age
GI tolerance | 1-120 days of age

OTHER OUTCOMES:
Influence on the microbial content of the stool | 3 - 4 times: 1-16 d, 4 w 16 w and 36 w
  Stool were collected to analyze the microbial content of certain bacteria upon enrollment and at the age of 4, 16. and 36 w Stool were collected and delivery to the lab in coolers within 12 h

CONTACTS AND LOCATIONS:
Overall Officials: Nehama Linder, M.D. Ph.D, Principal Investigator — Neonatology department, Rabin Medical center, Petach Tikva. Israel; Raanan Shamir, M.D. Ph.D., Principal Investigator — Institute of Gastroenterology Nutrition and Liver Diseases Schneider children medical center, Petach Tikva.; Kobi Shiff, M.D., Principal Investigator — Neonatology department, Laniado Hospital- Sanz Medical Center, Netanya, Israel.; Zvi Weizman, M.D. Ph.D, Principal Investigator — Department of Pediatrics, Soroka University Medical Center, Beer-Sheva, Israel.; Uri Rubenstein, M.D, Principal Investigator — clinic, 1 Yehuda Perach St., Natanya
Locations (1):
- Neonatology department, Laniado Hospital- Sanz Medical Center, ., Netanya, Israel